CLINICAL TRIAL: NCT04303364
Title: CARdiomyopathy in Type 2 DIAbetes Mellitus
Acronym: CARDIATEAM
Status: Recruiting | Type: Observational
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Collaborators: Consorcio Centro de Investigación Biomédica en Red (CIBER) (Other Government)
Responsible Party: Sponsor
Other Study IDs: C19-10
Record Dates: First submitted 2020-03-06; First posted 2020-03-11 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Cardiomyopathy, Diabetic
Keywords: Type2 Diabetes Mellitus; Heart Failure with preserved ejection fraction
MeSH Terms: conditions — Diabetic Cardiomyopathies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma EDTA, Serum, Paxgene RNA, Urine
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Subjects without T2DM and without HF
- Patients without T2DM and with HFpEF
- Patients with T2DM and without HFpEF
- Patients with T2DM and HFpEF
- Patients without T2DM and with hypertrophic cardiomyopathy
- Patients with T2DM and with hypertrophic cardiomyopathy

SUMMARY:
The objective of the CARDIATEAM clinical study is to assess the uniqueness of diabetic cardiomyopathy (DCM) relative to other forms of cardiomyopathy using unsupervised clustering approaches based on deep phenotyping (clinical, imaging and biological) information.

DETAILED DESCRIPTION:
CARDIATEAM study will address the uniqueness of DCM, and its progression towards heart failure (HF) with preserved ejection fraction (HFpEF) by recruiting a prospective CARDIATEAM cohort (n=1600 individuals) from existing cohorts using a defined set of selection criteria and will include type2-Diabetes mellitus (T2DM)and non-diabetic patients with a large spectrum of demographic, metabolic and cardiac clinical data. This will yield a wide range of T2DM - related phenotypes including common confounders such as BMI, smoking, age and blood pressure.

To clarify the phenotype of DCM and to differentiate it from the other forms of HF such as HFpEF or HCM, CARDIATEAM will perform unbiased clustering analysis from an in-depth phenotyping of these patients' populations

ELIGIBILITY:
Inclusion criteria

* Female or male, aged between ≥ 40 and ≤80 years
* Normal LVEF AND absence of akinetic segment assessed by echocardiography (i.e. LVEF≥50%)
* Patients diagnosed according to the specific diagnostic criteria of each disease (Cf. table below (definition criteria)). For each group, the diagnosis will be based on current accepted criteria:

  * HFpEF: left ventricular ejection fraction (LVEF) LVEF≥50% AND presence/or history of symptoms (e.g. breathlessness, ankle swelling and fatigue) or signs (e.g. elevated jugular venous pressure, pulmonary crackles and peripheral oedema) of heart failure AND significant diastolic dysfunction (left atrial volume index >34 mL/m2 or a LVMI ≥115 g/m2 for males and ≥95 g/m2 for female, E/e' ≥13 and e' <9 cm/s) OR NT-proBNP >125 pg/Ml
  * No HFpEF: LVEF≥50% AND absence of symptoms (e.g. breathlessness, ankle swelling and fatigue) or signs (e.g. elevated jugular venous pressure, pulmonary crackles and peripheral oedema) of heart failure
  * T2DM: HbA1c ≥ 6.5% (≥ 48 mmol/L) AND Fasting Plasma Glucose ≥7.0 mmol/L (≥126 mg/dL) or anti-diabetic treatment
  * Non T2DM: HbA1c < 6.5% AND Fasting Plasma Glucose <7.0 mmol/L without any anti-diabetic treatment including normoglycemic subjects
  * HCM: patients with non-obstructive HCM of sarcomeric cause (proven with common genetic cause) and with LV wall thickness ≥ 15 mm in one or more myocardial segments in the absence of abnormal afterload conditions.
* Suitable echocardiographic window
* Absence of history of coronary artery disease including history of myocardial ischaemia, myocardial infarction or percutaneous coronary intervention
* Absence of significant coronary artery disease (CAD) defined as:

  * the absence of coronary artery stenosis ≥50% on a cardiac computed tomography (CT) OR a coronary angiography OR normal Fractional Flow Reserve (FFR >0.80) OR
  * Coronary Artery Calcium score (CAC) <100 performed within the 48 months before inclusion
* Patient covered by a health insurance

Non-inclusion criteria:

* Diabetes mellitus other than type 2 (type 1, LADA, MODY, NODAT, etc.)
* Suboptimal echocardiographic window
* Significant valvular heart disease defined as severe aortic regurgitation or severe primary mitral regurgitation or aortic stenosis with a peak transvalvular velocity ≥3m/s or mitral stenosis with a mitral valve area < 1.5cm²
* Chronic atrial fibrillation or any significant arrhythmia at inclusion
* Renal insufficiency defined as eGFR<30 mL/min/1.73m²
* History of and candidate to bariatric surgery
* Obstructive hypertrophic cardiomyopathy (definition: maximal gradient at rest <30 mmHg)
* Hypertrophic cardiomyopathy due to a non-sarcomeric etiology, i.e. known infiltrative or storage disorder mimicking HCM such as Fabry disease or amyloidosis
* Life threatening comorbidities (i.e. history of or active cancer treated with chemotherapy or radiotherapy, end-stage heart failure, severe lung disease, cirrhosis)
* Pregnancy/Lactating mother
* Any condition which in the Investigator's opinion makes it undesirable for the subject to participate in the study or which would jeopardize compliance with the protocol
* Inability to understand the local language
* Individuals deprived of liberty
* Protected persons (under guardianship or curatorship)
* Contra-indication to CMR (please see CMR-SOP):
* Known hypersensitivity to gadolinium based product (including gadoteric acid and meglumine)
* Known COVID-19 symptomatic infection requiring hospitalization

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Since CARDIATEAM aims to assess the uniqueness of DCM, it will include a group of non-diabetic non-HFpEF individuals with diversified characteristics relating to obesity, glucose intolerance and hypertension. Consequently, CARDIATEAM cohort will recruit both non-diabetic and diabetic patients with a large spectrum of demographic, metabolic and cardiac (heart failure vs. no heart failure) clinical data.
Sampling Method: Non-Probability Sample
Enrollment: 1600 (Estimated)
Dates: Start 2020-10-02 (Actual); Primary Completion 2028-04-01 (Estimated); Study Completion 2028-04-01 (Estimated)

PRIMARY OUTCOMES:
Assess the uniqueness of diabetic cardiomyopathy (DCM) relative to other forms of cardiomyopathy | 3 years
  Use of unsupervised clustering approaches based on deep phenotyping (clinical, imaging and biological) information

SECONDARY OUTCOMES:
Identify the best clinical, biological, imaging and multi-OMICs predictors belonging to each identified cluster | 4 years
  Specific focus on cluster(s) relating to a putative diabetic cardiomyopathy comparatively to other clusters [diagnostic perspective]
Assess prospective health outcomes (i.e. overall mortality, cardiovascular events and cardiac function) in the diabetic cardiomyopathy cluster identified | 5 years
  Compare them to those from the other clusters and pre-defined patient groups [prognostic perspective]
Explore the pathophysiological and potentially causal pathways characterizing diabetic cardiomyopathy | 5 years
  Better understand the underlying mechanisms responsible for establishment and progression of disease, based on OMICs data and causal inference modeling

CONTACTS AND LOCATIONS:
Overall Officials: Geneviève DERUMEAUX, MD, PhD, Principal Investigator — Henri Mondor University Hospital
Locations (17):
- France (7):
  - Hopital Louis Pradel, Bron
  - Cardiology Outpatient Department at Hôpital Henri Mondor., Créteil
  - Centre Hospitalier Universitaire Grenoble Alpes, Grenoble
  - department of diabetology and nutrition, APHM, Marseille
  - Hôpital CHU- Nantes, Nantes
  - Diabetology department, Cochin Institute, Paris
  - Diabetology departement, Lariboisière Hospital, Paris
- Germany (2):
  - University Hospital Aachen, Aachen
  - University Hospital Heidelberg, Heidelberg
- Netherlands (4):
  - Amsterdam UMC, Amsterdam
  - University Medical Center Groningen (UMCG), Cardiology/Cardio Research, Groningen
  - Academisch ziekenhuis Maastricht, Cardiology, Maastricht
  - UMC Utrecht, Cardiology (DHL), Utrecht
- Spain (3):
  - Hospital Vall Hebrón, Barcelona
  - Institut D'Investigacions Biomedica August Pi I Sunyer (IDIBAPS), Barcelona
  - Hospital Gregorio Marañón, Madrid
- University of Dundee, Div of Molecular&Clinical Medicine, Dundee, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided